CLINICAL TRIAL: NCT01595659
Title: Influence of Alcohol and Peer Passengers on Risky Driving Behavior in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie Claude Ouimet, Associate professor, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MOP-111034
Record Dates: First submitted 2012-05-05; First posted 2012-05-10 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Accidents, Traffic
Keywords: Risk; Young drivers; Alcohol; Passengers; Gender
MeSH Terms: conditions — Coitus | interventions — nuclear passenger protein-1, S pombe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no alcohol and passenger (Placebo Comparator): Blood alcohol concentration (BAC) = 0.00% and risk accepting or averse passenger
  Interventions: Behavioral: Passenger
- low alcohol dose and passenger (Experimental): BAC = 0.02% and risk accepting or averse passenger
  Interventions: Behavioral: Passenger
- moderate alcohol dose and passenger (Experimental): BAC = 0.05% and risk accepting or averse passenger
  Interventions: Behavioral: Passenger

INTERVENTIONS:
Behavioral: Passenger — Driving with risk accepting or risk averse passenger

SUMMARY:
Among the many risk factors that contribute to young drivers' crash involvement, two are critical: peer passenger presence, which is unique to young drivers, and the influence of alcohol, a universal risk for drivers but one against which young drivers are most susceptible. Clarification of how passenger presence interacts with alcohol consumption to increase risk is needed. The impact of experimentally manipulated passenger characteristics and alcohol quantity on risky driving is observed using driving simulation and a random assignment experimental design with a sample of 18-21 year old male and female drivers.

ELIGIBILITY:
Inclusion Criteria:

* being 18 to 21 years of age (18 years old is the legal age for alcohol consumption in the province of Quebec)
* past experirence with drinking at least 2 alcoholic beverages in one episode
* having a provisional driving license
* driving in the past 3 months

Exclusion Criteria:

* health problem that contraindicates participation
* pregnant or breastfeeding
* signs of problem drinking
* positive BAC or recent drug use measured at arrival

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-06-03 (Actual)

PRIMARY OUTCOMES:
Risky driving in a simulator | within 1 hr after alcohol dose

CONTACTS AND LOCATIONS:
Overall Officials: Marie Claude Ouimet, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Longueuil, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No